CLINICAL TRIAL: NCT03582657
Title: Multicenter, Prospective, Observational Study on the Performance and Safety Use of the Dental Implant "KONTACT N" in the Current Clinical Practice
Brief Title: Performance and Safety Use of the Nanostructured Titanium Dental Implant "KONTACT N"
Status: Completed | Type: Observational
Sponsor: Biotech Dental (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-A00194-51
Record Dates: First submitted 2018-06-15; First posted 2018-07-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Dental Implant; Dental Restoration; Edentulous Alveolar Ridge; Implant-supported Fixed Prosthesis
Keywords: nanostructured-implant; titanium implant; nano-roughness surface; hydrophilic surface; KONTACT N; BIOTECH DENTAL
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: dental implant (KONTACT N) — Implant-supported prosthetic restoration
  Other Names: KONTACT N; BIOTECH DENTAL

SUMMARY:
A multicenter prospective observational study in which aim is to illustrate the clinical outcome of dental implants "Kontact N"; and the effects of its nanostructured surface on the osseointegration and secondary stability without increasing the rate of peri-implantitis. All the enrolled patients will be eligible for one or multiple implant-supported fixed restoration(s) according to the routine clinical practice and the manufacturer's instruction for use.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous patient (partially or completely AND formerly, recently or just before implantation) requiring the placement of one (or more) dental implant (s) in maxillary or mandibular
* Age ≥ 18 years
* Good general health (ASA score between [1-2])
* Sufficient bone volume and quality (with or without bone graft) to support the implant
* Non-opposition of the patient for the collection of his medical data as part of the study (delivery of a patient's sheet)

Exclusion Criteria:

1. Poor oral hygiene
2. Bruxism, parafunctional habits, occlusion disorders and / or temporomandibular joints
3. Infections and oral inflammation such as periodontitis, gingivitis
4. Patient with metabolic disorders (eg diabetes mellitus) or bone disease that may compromise peri-implant tissue healing
5. Heavy smoker (> 10 cigarettes / day)
6. Patient with a pathology or immunosuppressive therapy such as chemotherapy, radiotherapy
7. Patient on prolonged steroid therapy
8. Titanium / titanium alloy allergy
9. Alcohol or drug abuse
10. Pregnant woman (or likely to be pregnant); or breastfeeding
11. Difficulty of medical follow-up patients with geographical, social or psychological constraints
12. Persons deprived of liberty or guardianship
13. Involuntary / patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who is eligible and planned for an implant-supported prosthetic restoration following the instructions for use of the KONTACT N implant and who meets the inclusion / exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Implant success rate | up to 12 months post-implantation
  Rate of implants still in function up to 12 months post-implantation and which fulfill all the predefined success criteria in the protocol.
Peri-implantitis rate | 12 months post-implantation
  Peri-implantitis is an inflammatory process affecting the tissues around the implant and causing loss of bone support (diagnosed by radiographic and clinical assessment).
Mean osseointegration period | From the implantation up to 12 months
  Period from which a direct structural and functional junction can be observed between the remodeled living bone and the implant surface (by clinical and radiographic assessment).

CONTACTS AND LOCATIONS:
Overall Officials: KHOURY, Dr, Principal Investigator
Locations (1):
- Dr KHOURY Elias, Paris, France

IPD SHARING:
Plan to Share IPD: No